CLINICAL TRIAL: NCT00821340
Title: Phase I Trial of Ocular Subretinal Injection of a Recombinant Adeno-Associated Virus (rAAV2-hRPE65) Gene Vector to Patients With Retinal Disease Due to RPE65 Mutations
Brief Title: Clinical Trial of Gene Therapy for Leber Congenital Amaurosis Caused by RPE65 Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPE65-HMO-CTIL
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2010-02

CONDITIONS: Leber Congenital Amaurosis
Keywords: Leber congenital amaurosis; LCA; RPE65; RPE65-associated Leber congenital amaurosis; Retinal disease due to RPE65 mutations
MeSH Terms: conditions — Leber Congenital Amaurosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rAAV2-hRPE65 (Experimental)
  Interventions: Genetic: rAAV2-hRPE65

INTERVENTIONS:
Genetic: rAAV2-hRPE65 — Uniocular subretinal injections; relative doses: Cohort 1 - basic (lowest) viral dose; Cohort 2 - higher (1.5 times basic) viral dose; Cohort 3 - patients 8-17 years of age will receive basic viral dose; patients 18 years of age and over will receive higher dose;

SUMMARY:
The purpose of this clinical trial is to examine the safety of gene therapy for Lebers Congenital Amaurosis (LCA) caused by RPE65 mutations using a recombinant adeno-associated virus serotype 2 (rAAV2) vector carrying the human RPE65 (hRPE65) gene. Recently, three independent short-term gene therapy studies in humans with LCA due to RPE65 mutations were published, suggesting that subretinal delivery of rAAV virus carrying the RPE65 gene is safe. As a secondary outcome, improvement in visual function was observed in seven of the first nine treated patients. The proposed study is a similar open label, Phase I clinical trial of uniocular subretinal rAAV2-hRPE65 administration to individuals with RPE65-associated retinal disease. Two cohorts of three subjects each and one cohort of four subjects will be included in this trial. Cohort 1 and 2 will consist of individuals 18 years of age and older and Cohorts 3 will consist of individuals 8 years of age and older. In cohort 2, a larger volume of vector will be administered. Enrollment in Cohort 3 will begin only after confirming the safety of rAAV2-hRPE65 administration in the older group of participants.

ELIGIBILITY:
Inclusion Criteria:

* Retinal disease caused by homozygous or compound heterozygote RPE65 mutations;
* Clinical diagnosis of Leber congenital amaurosis (LCA) with severely impaired visual and retinal function, and best corrected visual acuity of 20/50 or worse in the study eye;
* Ability to perform tests of visual and retinal function;
* Good general health;
* Ability to comply with research procedures;
* Specific for Cohort 1 and 2: 18 years of age and older;
* Specific for Cohort 3: Over 8 years of age;

Exclusion Criteria:

* Immune deficiency or use of immunosuppressive medications;
* Pre-existing eye conditions that would preclude the planned surgery or interfere with the interpretation of study endpoints (for example, glaucoma or ocular media opacities);
* Complicating systemic diseases;
* Impaired coagulation or use of anti-platelet agents within 7 days prior to study agent administration;
* Pregnancy or breastfeeding;
* Individuals (males and females) of childbearing potential who are unwilling to use effective contraception for 1 year following agent administration and barrier contraception for 3 months following agent administration;
* Any other condition that would prevent a subject from completing follow-up examinations during the course of the study;
* Any other condition that, in the opinion of the investigator, makes the subject unsuitable for the study;
* Current or recent participation in any other research protocol involving investigational agents or therapies, including recent (within past 6 months) receipt of an investigational biologic therapeutic agent.

Subjects will not be excluded based on their gender, race or ethnicity.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is ocular and systemic safety of the treatment. | 3 years

SECONDARY OUTCOMES:
Visual function, as quantified before and after vector administration. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Banin, MD, PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acland GM, Aguirre GD, Bennett J, Aleman TS, Cideciyan AV, Bennicelli J, Dejneka NS, Pearce-Kelling SE, Maguire AM, Palczewski K, Hauswirth WW, Jacobson SG. Long-term restoration of rod and cone vision by single dose rAAV-mediated gene transfer to the retina in a canine model of childhood blindness. Mol Ther. 2005 Dec;12(6):1072-82. doi: 10.1016/j.ymthe.2005.08.008. Epub 2005 Oct 14. PMID 16226919
- [Background] Bainbridge JW, Smith AJ, Barker SS, Robbie S, Henderson R, Balaggan K, Viswanathan A, Holder GE, Stockman A, Tyler N, Petersen-Jones S, Bhattacharya SS, Thrasher AJ, Fitzke FW, Carter BJ, Rubin GS, Moore AT, Ali RR. Effect of gene therapy on visual function in Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2231-9. doi: 10.1056/NEJMoa0802268. Epub 2008 Apr 27. PMID 18441371
- [Background] Maguire AM, Simonelli F, Pierce EA, Pugh EN Jr, Mingozzi F, Bennicelli J, Banfi S, Marshall KA, Testa F, Surace EM, Rossi S, Lyubarsky A, Arruda VR, Konkle B, Stone E, Sun J, Jacobs J, Dell'Osso L, Hertle R, Ma JX, Redmond TM, Zhu X, Hauck B, Zelenaia O, Shindler KS, Maguire MG, Wright JF, Volpe NJ, McDonnell JW, Auricchio A, High KA, Bennett J. Safety and efficacy of gene transfer for Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2240-8. doi: 10.1056/NEJMoa0802315. Epub 2008 Apr 27. PMID 18441370
- [Background] Miller JW. Preliminary results of gene therapy for retinal degeneration. N Engl J Med. 2008 May 22;358(21):2282-4. doi: 10.1056/NEJMe0803081. Epub 2008 Apr 27. No abstract available. PMID 18441372
- [Background] Hauswirth WW, Aleman TS, Kaushal S, Cideciyan AV, Schwartz SB, Wang L, Conlon TJ, Boye SL, Flotte TR, Byrne BJ, Jacobson SG. Treatment of leber congenital amaurosis due to RPE65 mutations by ocular subretinal injection of adeno-associated virus gene vector: short-term results of a phase I trial. Hum Gene Ther. 2008 Oct;19(10):979-90. doi: 10.1089/hum.2008.107. PMID 18774912
- [Background] Cideciyan AV, Aleman TS, Boye SL, Schwartz SB, Kaushal S, Roman AJ, Pang JJ, Sumaroka A, Windsor EA, Wilson JM, Flotte TR, Fishman GA, Heon E, Stone EM, Byrne BJ, Jacobson SG, Hauswirth WW. Human gene therapy for RPE65 isomerase deficiency activates the retinoid cycle of vision but with slow rod kinetics. Proc Natl Acad Sci U S A. 2008 Sep 30;105(39):15112-7. doi: 10.1073/pnas.0807027105. Epub 2008 Sep 22. PMID 18809924